CLINICAL TRIAL: NCT03280927
Title: A Multicenter, Open-label, Non-controlled, Single-arm Phase IV Clinical Trial to Evaluate the Efficacy and Safety of Jublia® in Mild to Moderate Toenail Onychomycosis
Brief Title: Phase IV Clinical Trial to Evaluate the Efficacy and Safety of Jublia® in Mild to Moderate Toenail Onychomycosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JBL_OM_IV
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Mild to Moderate Onychomycosis Due to Dermatophyte
Keywords: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — efinaconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jublia® (Experimental)
  Interventions: Drug: Jublia®

INTERVENTIONS:
Drug: Jublia® — Jublia® topical solution

SUMMARY:
The antifungal efficacy and safety of Jublia® topical solution will be assessed through an administration for 48 weeks to patients diagnosed with a mild or moderate onychomycosis due to dermatophyte.

DETAILED DESCRIPTION:
Evaluate anti-fungal activity and safety of efinaconazole in patients with mild to moderate toenail onychomycosis caused by dermatophytes that received a 48-week administration of efinaconazole.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects of ages in the range over 19.
* The subjects diagnosed with onychomycosis in up to 6 toenails at least

  1 great toenail woth no fingernails
* The subjects diagnosed with a mild to moderate onychomycosis (20% to 50% of surface of target nail without nail matrix infection or dermatophytoma)
* The subjects having target nails less than 3mm in thickness and over 3mm in length
* Positive indication on KOH Direct Microscopic Inspection on target nail
* Positive dermatophyte or dermatophyte/candida on Fungi Cultivation Inspection on target nail
* The subjects completely understood the clinical trial through detailed explanation presented, determined to participate in the clinical trial spontaneously, and agreed to observe precautions suggested thereby through written consent.

Exclusion Criteria:

* The subjects suffering other diseases that may cause nail abnormalities or are supposed to be affecting the assessment of the efficacy of study agent by the judgment of investigators
* The subjects having a case history of hypersensitivity reaction to the component of Jublia® topical solution or Azole derivatives.
* The pregnant, lactating, or fertile woman free from pertinent contraception

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Completely cured subjects | 52 weeks
  The ratio of completely cured subjects

SECONDARY OUTCOMES:
Complete or almost complete cure rates | 52 weeks
  The ratio of subjects showing less than 5% of infection area
Mycologic cure rates | 52 weeks
  Negative results from both the KOH Direct Microscopic Inspection and Fungi Cultivation Inspection.
Clinical efficacy rates | 52 weeks
  The ratio of subjects affected target nail area less than 10%

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea